CLINICAL TRIAL: NCT02604212
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Multi-dose Study to Determine the Depth of Hepatitis B Surface Antigen (HBsAg) Reduction Following Intravenous ARC-520 in Combination With Entecavir or Tenofovir in Patients With HBeAg Positive, Chronic Hepatitis B Virus (HBV) Infection
Brief Title: A Multi-dose Study of ARC-520 in Patients With Hepatitis B 'e' Antigen (HBeAg) Positive, Chronic Hepatitis B Virus Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to discontinue trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Heparc-2003; 2014-004751-31 (EudraCT Number)
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — ARC-520; entecavir; Histamine Antagonists; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Low Dose Comparator (Placebo Comparator): Placebo (low dose comparator) once every 4 weeks for 4 doses, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day)
  Interventions: Other: Placebo; Drug: entecavir; Drug: antihistamine; Drug: tenofovir
- Placebo High Dose Comparator (Placebo Comparator): Placebo (high dose comparator) once every 4 weeks for 4 doses, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day)
  Interventions: Other: Placebo; Drug: entecavir; Drug: antihistamine; Drug: tenofovir
- ARC-520 1.0 mg/kg (Experimental): Low dose (1.0 mg/kg) ARC-520 once every 4 weeks for 4 doses, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day)
  Interventions: Drug: ARC-520; Drug: entecavir; Drug: antihistamine; Drug: tenofovir
- ARC-520 2.0 mg/kg (Experimental): High dose (2.0 mg/kg) ARC-520 once every 4 weeks for 4 doses, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day)
  Interventions: Drug: ARC-520; Drug: entecavir; Drug: antihistamine; Drug: tenofovir

INTERVENTIONS:
Drug: ARC-520
  Arms: ARC-520 1.0 mg/kg; ARC-520 2.0 mg/kg
Other: Placebo
  Arms: Placebo High Dose Comparator; Placebo Low Dose Comparator
Drug: entecavir — All participants will take entecavir or tenofovir throughout the study. Participants will be instructed to take their medication daily.
Drug: antihistamine — All participants will be pretreated with an oral antihistamine. The antihistamine used should in general be an H1>H2 receptor blocker and would include diphenhydramine 50 mg, cetirizine 10 mg, chlorpheniramine 8 mg or hydroxyzine 50 mg. The Investigator is free to choose any of these antihistamines available locally and consistent with their country's Marketing Authorisation.
Drug: tenofovir — All participants will take entecavir or tenofovir throughout the study. Participants will be instructed to take their medication daily.

SUMMARY:
Patients with HBeAG positive, chronic HBV infection will receive either ARC-520 or placebo in combination with entecavir or tenofovir, and be evaluated for safety and efficacy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, multi-dose study of ARC-520 in combination with entecavir or tenofovir administered to patients with HBeAg positive and immune active chronic HBV infection Eligible patients who have signed an Ethics Committee - approved informed consent, will be enrolled and will receive ARC-520 or placebo in combination with entecavir or tenofovir. The study will enroll up to a total of 90 eligible chronic HBV infected patients. Patients will undergo the following evaluations at regular intervals during the study: medical history, physical examinations, vital sign measurements (blood pressure, heart rate, respiratory rate and temperature), weight, adverse events assessment (AEs), 12 lead electrocardiograms (ECGs), liver fibrosis testing, concomitant medication assessment, blood sample collection for hematology, coagulation, chemistry, lactate, Pharmacokinetic (PK) measures (in a subset of patients), exploratory Pharmacodynamic (PD) measures, urinalysis, HBV serology, Follicle Stimulating Hormone (FSH) testing (post-menopausal females) and pregnancy testing for females of childbearing potential. Clinically significant changes including AEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the patient is lost to follow-up. For each patient the duration of the study is approximately 33 weeks from screening to the Day 169 follow-up visit. For patients enrolling into a planned extension study, the total duration of this study is approximately 25 weeks from screening to Day 113 end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age.
* Written informed consent.
* No clinically significant abnormalities at screening/pre-dose 12-lead ECG assessment.
* No new abnormal finding of clinical relevance at the screening evaluation.
* Diagnosis of HBeAg positive, immune active, chronic HBV infection.
* > 2months of continuous treatment with daily, oral entecavir or tenofovir.
* Willingness to continue taking entecavir or tenofovir throughout the study.
* Must use 2 effective methods of contraception (double barrier contraception or hormonal contraceptive along with a barrier contraceptive) (both male and female partners).

Exclusion Criteria:

* Pregnant or lactating
* Acute signs of hepatitis/other infection within 4 weeks of screening.
* Antiviral therapy other than entecavir or tenofovir within 3 months of screening.
* Prior treatment with interferon in the last 3 years.
* Use within the last 6 months or anticipated requirement for anticoagulants, corticosteroids, immunomodulators, or immunosuppressants.
* Use of prescription medication within 14 days prior to treatment administration except: topical products without systemic absorption, statins (except rosuvastatin), hypertension medications, or hormonal contraceptives.
* Depot injection or implant of any drug within 3 months prior to treatment administration, except injectable/implantable birth control.
* Diagnosis of diabetes mellitus.
* History of autoimmune disease especially autoimmune hepatitis.
* Human immunodeficiency virus (HIV) infection.
* Sero-positive for Hepatitis C Virus (HCV), and/or a history of delta virus hepatitis.
* Hypertension defined as blood pressure > 150/100 mmHg.
* History of cardiac rhythm disturbances.
* Family history or congenital long QT syndrome, Brugada syndrome or unexplained sudden cardiac death.
* Symptomatic heart failure, unstable angina, myocardial infarction, severe cardiovascular disease within 6 months prior to study entry.
* History of malignancy except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer.
* Has had a major surgery within 3 months of screening.
* History of alcohol and/or drug abuse < 12 months from screening.
* Regular uses of alcohol within 6 months prior to screening (ie, more than 14 units of alcohol per week).
* Evidence of severe systemic acute inflammation, sepsis, or hemolysis.
* Diagnosed with a significant psychiatric disorder.
* Use of recreational drugs, such as marijuana, within 3 months prior to screening.
* Use of drugs such as cocaine, phencyclidine (PCP), and methamphetamines, within 1 year prior to screening.
* History of allergy to bee sting.
* Use of investigational agents or devices within 30 days prior to planned study dosing or current participation in an investigational study.
* Clinically significant history or presence of any gastrointestinal pathology, unresolved gastrointestinal symptoms, liver or kidney disease.
* Presence of cholangitis, cholecystitis, cholestasis, or duct obstruction.
* Clinically significant history or presence of poorly controlled/uncontrolled systemic disease.
* History of fever within 2 weeks of screening.
* Immunized with a live attenuated vaccine within 7 days prior to dosing or planned vaccination (excluding flu vaccine by injection).
* Presence of any medical or psychiatric condition or social situation that impacts compliance or results in additional safety risk.
* Participated in excessive exercise/physical activity within 7 days of screening or planned during the trial.
* History of coagulopathy/stroke within past 6 months, and/or concurrent anticoagulant medication(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- China (2):
  - Research Site 1, Hong Kong
  - Research Site 2, Hong Kong
- Germany (9):
  - Research Site 11, Frankfurt
  - Research Site 9, Hamburg
  - Research Site 8, Hanover
  - Research Site 10, Leipzig
  - Research Site 4, Leipzig
  - Research Site 5, München
  - Research Site 3, Tübingen
  - Research Site 6, Ulm
  - Research Site 7, Würzburg
- South Korea (5):
  - Research Site 13, Busan
  - Research Site 15, Incheon
  - Research Site 14, Seoul
  - Research Site 16, Seoul
  - Research Site 12, Yangsan-si Gyeongnam

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Low Dose Comparator | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Started | 6 | 5 | 10 | 11
Completed | 4 | 4 | 6 | 8
Not Completed | 2 | 1 | 4 | 3
Not completed — Study Terminated by Sponsor | 2 | 1 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Low Dose Comparator | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg | Total
Number analyzed (Participants) | 6 | 5 | 10 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (9.54) | 45.0 (10.68) | 42.1 (12.57) | 41.6 (12.05) | 42.0 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 6 | 10
  Male | 3 | 4 | 10 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Quantitative Hepatitis B Surface Antigen (Log qHBsAg) at Day 113
Description: Change From Baseline in log qHBsAg at Day 113 in response to multiple doses of ARC-520 versus placebo, using a a mixed effect model for repeated measures (MMRM). Includes parameter baseline as a continuous covariate, and treatment and visit as fixed factors, interaction of treatment and visit, and interaction of parameter baseline and visit.
Time Frame: Baseline, Day 113
Population: Intent to treat population: all participants who received at least 1 dose of study drug and had valid qHBsAg values at baseline and at least one time point on or after the Day 15 visit.
Measure: Least Squares Mean (Standard Error); unit: log IU/mL
Groups:
- Placebo: Placebo (low or high dose comparator) once every 4 weeks for 4 doses, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day)
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 8
log IU/mL | -0.104 (0.073) | -0.146 (0.065) | -0.542 (0.061)
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Test type: Superiority; p = 0.6815, MMRM; LS Mean Difference = -0.042, 95% CI 2-sided [-0.243 to 0.159], Standard Error of Mean 0.102
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Test type: Superiority; p < .0001, MMRM; LS Mean Difference = -0.438, 95% CI 2-sided [-0.638 to -0.237], Standard Error of Mean 0.101
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Test type: Superiority; p < .0001, MMRM; LS Mean Difference = -0.396, 95% CI 2-sided [-0.569 to -0.223], Standard Error of Mean 0.088

2. Secondary Outcome: Change From Baseline in Log qHBsAg Over Time
Description: Change From Baseline in log qHBsAg up to Day 99 in response to multiple doses of ARC-520 versus placebo, using a a mixed effect model for repeated measures (MMRM). Includes parameter baseline as a continuous covariate, and treatment and visit as fixed factors, interaction of treatment and visit, and interaction of parameter baseline and visit.
Time Frame: Baseline, Days 15, 29, 43, 57, 71, 85, 99
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Groups:
- Placebo: Placebo (low dose or high dose comparator) once every 4 weeks for 4 doses, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day)
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 10 | 10 | 10
log IU/mL
  Day 15 | 3.734 (0.519) | 3.069 (0.654) | 3.000 (0.411)
  Day 29: number analyzed (Participants) | 9 | 10 | 10
  Day 29 | 3.692 (0.588) | 3.148 (0.658) | 3.027 (0.395)
  Day 43: number analyzed (Participants) | 8 | 9 | 10
  Day 43 | 3.812 (0.463) | 3.097 (0.664) | 2.893 (0.436)
  Day 57: number analyzed (Participants) | 7 | 9 | 10
  Day 57 | 3.793 (0.507) | 3.148 (0.651) | 2.882 (0.437)
  Day 71: number analyzed (Participants) | 7 | 9 | 9
  Day 71 | 3.756 (0.489) | 3.088 (0.626) | 2.714 (0.477)
  Day 85: number analyzed (Participants) | 7 | 7 | 8
  Day 85 | 3.743 (0.543) | 3.198 (0.610) | 2.698 (0.466)
  Day 99: number analyzed (Participants) | 7 | 6 | 8
  Day 99 | 3.767 (0.541) | 3.048 (0.593) | 2.606 (0.477)
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Day 15; Test type: Superiority; p = 0.0131, MMRM; LS Mean Difference = -0.208, 95% CI 2-sided [-0.372 to -0.044], Standard Error of Mean 0.083
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Day 15; Test type: Superiority; p = 0.0036, MMRM; LS Mean Difference = -0.247, 95% CI 2-sided [-0.412 to -0.082], Standard Error of Mean 0.084
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Day 15; Test type: Superiority; p = 0.6136, MMRM; LS Mean Difference = -0.039, 95% CI 2-sided [-0.192 to 0.113], Standard Error of Mean 0.077
Statistical Analysis 4: Comparison: Placebo vs ARC-520 1.0 mg/kg; Day 29; Test type: Superiority; p = 0.3104, MMRM; LS Mean Difference = -0.085, 95% CI 2-sided [-0.249 to 0.080], Standard Error of Mean 0.083
Statistical Analysis 5: Comparison: Placebo vs ARC-520 2.0 mg/kg; Day 29; Test type: Superiority; p = 0.0401, MMRM; LS Mean Difference = -0.174, 95% CI 2-sided [-0.340 to -0.008], Standard Error of Mean 0.084
Statistical Analysis 6: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Day 29; Test type: Superiority; p = 0.2494, MMRM; LS Mean Difference = -0.089, 95% CI 2-sided [-0.242 to 0.063], Standard Error of Mean 0.077
Statistical Analysis 7: Comparison: Placebo vs ARC-520 1.0 mg/kg; Day 43; Test type: Superiority; p = 0.0149, MMRM; LS Mean Difference = -0.211, 95% CI 2-sided [-0.380 to -0.042], Standard Error of Mean 0.085
Statistical Analysis 8: Comparison: Placebo vs ARC-520 2.0 mg/kg; Day 43; Test type: Superiority; p = 0.0003, MMRM; LS Mean Difference = -0.319, 95% CI 2-sided [-0.489 to -0.149], Standard Error of Mean 0.086
Statistical Analysis 9: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Day 29; Test type: Superiority; p = 0.1655, MMRM; LS Mean Difference = -0.108, 95% CI 2-sided [-0.262 to 0.045], Standard Error of Mean 0.078
Statistical Analysis 10: Comparison: Placebo vs ARC-520 1.0 mg/kg; Day 57; Test type: Superiority; p = 0.0889, MMRM; LS Mean Difference = -0.150, 95% CI 2-sided [-0.324 to 0.023], Standard Error of Mean 0.088
Statistical Analysis 11: Comparison: Placebo vs ARC-520 2.0 mg/kg; Day 57; Test type: Superiority; p = 0.0004, MMRM; LS Mean Difference = -0.322, 95% CI 2-sided [-0.497 to -0.147], Standard Error of Mean 0.088
Statistical Analysis 12: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Day 57; Test type: Superiority; p = 0.0298, MMRM; LS Mean Difference = -0.172, 95% CI 2-sided [-0.326 to -0.017], Standard Error of Mean 0.078
Statistical Analysis 13: Comparison: Placebo vs ARC-520 1.0 mg/kg; Day 71; Test type: Superiority; p = 0.0415, MMRM; LS Mean Difference = -0.184, 95% CI 2-sided [-0.361 to -0.007], Standard Error of Mean 0.089
Statistical Analysis 14: Comparison: Placebo vs ARC-520 2.0 mg/kg; Day 71; Test type: Superiority; p < .0001, MMRM; LS Mean Difference = -0.441, 95% CI 2-sided [-0.620 to -0.261], Standard Error of Mean 0.091
Statistical Analysis 15: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Day 71; Test type: Superiority; p = 0.0015, MMRM; LS Mean Difference = -0.257, 95% CI 2-sided [-0.413 to -0.100], Standard Error of Mean 0.079
Statistical Analysis 16: Comparison: Placebo vs ARC-520 1.0 mg/kg; Day 85; Test type: Superiority; p = 0.3510, MMRM; LS Mean Difference = -0.086, 95% CI 2-sided [-0.268 to 0.096], Standard Error of Mean 0.092
Statistical Analysis 17: Comparison: Placebo vs ARC-520 2.0 mg/kg; Day 85; Test type: Superiority; p < .0001, MMRM; LS Mean Difference = -0.404, 95% CI 2-sided [-0.590 to -0.219], Standard Error of Mean 0.094
Statistical Analysis 18: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Day 85; Test type: Superiority; p = 0.0002, MMRM; LS Mean Difference = -0.318, 95% CI 2-sided [-0.481 to -0.156], Standard Error of Mean 0.082
Statistical Analysis 19: Comparison: Placebo vs ARC-520 1.0 mg/kg; Day 99; Test type: Superiority; p = 0.1198, MMRM; LS Mean Difference = -0.151, 95% CI 2-sided [-0.341 to 0.040], Standard Error of Mean 0.096
Statistical Analysis 20: Comparison: Placebo vs ARC-520 2.0 mg/kg; Day 99; Test type: Superiority; p < .0001, MMRM; LS Mean Difference = -0.516, 95% CI 2-sided [-0.708 to -0.325], Standard Error of Mean 0.097
Statistical Analysis 21: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Day 99; Test type: Superiority; p < .0001, MMRM; LS Mean Difference = -0.366, 95% CI 2-sided [-0.535 to -0.197], Standard Error of Mean 0.085

3. Secondary Outcome: Change From Baseline at Day 15 in Log qHBsAg, by Category
Description: Change in log qHBsAg from baseline, categorized into the following groups: no decrease, decrease > 0 to < 0.5 log IU/mL; decrease 0.5 to 1.0 log IU/mL; decrease > 1.0 log IU/mL, tabulated by dose and treatment for each visit.
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 10 | 10 | 10
log IU/mL
  No Decrease: number analyzed (Participants) | 4 | 0 | 2
  No Decrease | 0.026 (0.015) |  | 0.032 (0.035)
  Decrease > 0 to < 0.5 log IU/mL: number analyzed (Participants) | 6 | 9 | 7
  Decrease > 0 to < 0.5 log IU/mL | -0.035 (0.014) | -0.153 (0.144) | -0.266 (0.192)
  Decrease 0.5 to 1.0 log IU/mL: number analyzed (Participants) | 0 | 1 | 1
  Decrease 0.5 to 1.0 log IU/mL |  | -0.707 (NA) — 1 participant analyzed | -0.666 (NA) — 1 participant analyzed
  Decrease > 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Test type: Superiority; p = 0.0867, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.6285, Fisher Exact
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.7214, Fisher Exact

4. Secondary Outcome: Change From Baseline at Day 29 in Log qHBsAg, by Category
Description: as for outcome 3
Time Frame: Baseline, Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 9 | 10 | 10
log IU/mL
  No Decrease: number analyzed (Participants) | 4 | 0 | 1
  No Decrease | 0.048 (0.043) |  | 0.064 (NA) — 1 participant analyzed
  Decrease > 0 to < 0.5 log IU/mL: number analyzed (Participants) | 5 | 10 | 10
  Decrease > 0 to < 0.5 log IU/mL | -0.084 (0.078) | -0.129 (0.083) | -0.251 (0.190)
  Decrease 0.5 to 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 0
  Decrease > 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Test type: Superiority; p = 0.0325, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.1409, Fisher Exact
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 1.0000, Fisher Exact

5. Secondary Outcome: Change From Baseline at Day 43 in Log qHBsAg, by Category
Description: as for outcome 3
Time Frame: Baseline, Day 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 8 | 9 | 10
log IU/mL
  No Decrease: number analyzed (Participants) | 3 | 0 | 1
  No Decrease | 0.022 (0.012) |  | 0.017 (NA) — 1 participant analyzed
  1 participant analyDecrease > 0 to < 0.5 log IU/mL: number analyzed (Participants) | 5 | 9 | 6
  1 participant analyDecrease > 0 to < 0.5 log IU/mL | -0.050 (0.051) | -0.226 (0.077) | -0.275 (0.137)
  Decrease 0.5 to 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 3
  Decrease 0.5 to 1.0 log IU/mL |  |  | -0.633 (0.141)
  Decrease > 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Test type: Superiority; p = 0.0824, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.2217, Fisher Exact
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.1409, Fisher Exact

6. Secondary Outcome: Change From Baseline at Day 57 in Log qHBsAg, by Category
Description: as for outcome 3
Time Frame: Baseline, Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 7 | 9 | 10
log IU/mL
  No Decrease: number analyzed (Participants) | 3 | 0 | 0
  No Decrease | 0.027 (0.012) |  |
  1 participant analyDecrease > 0 to < 0.5 log IU/mL: number analyzed (Participants) | 4 | 9 | 7
  1 participant analyDecrease > 0 to < 0.5 log IU/mL | -0.067 (0.072) | -0.176 (0.049) | -0.276 (0.156)
  Decrease 0.5 to 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 3
  Decrease 0.5 to 1.0 log IU/mL |  |  | -0.571 (0.060)
  Decrease > 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Test type: Superiority; p = 0.0625, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.0684, Fisher Exact
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.2105, Fisher Exact

7. Secondary Outcome: Change From Baseline at Day 71 in Log qHBsAg, by Category
Description: as for outcome 3
Time Frame: Baseline, Day 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 7 | 9 | 9
log IU/mL
  No Decrease: number analyzed (Participants) | 2 | 0 | 0
  No Decrease | 0.011 (0.012) |  |
  1 participant analyDecrease > 0 to < 0.5 log IU/mL: number analyzed (Participants) | 5 | 9 | 4
  1 participant analyDecrease > 0 to < 0.5 log IU/mL | -0.094 (0.079) | -0.235 (0.086) | -0.296 (0.119)
  Decrease 0.5 to 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 5
  Decrease 0.5 to 1.0 log IU/mL |  |  | -0.662 (0.140)
  Decrease > 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Test type: Superiority; p = 0.1750, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.0229, Fisher Exact
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.0294, Fisher Exact

8. Secondary Outcome: Change From Baseline at Day 85 in Log qHBsAg, by Category
Description: as for outcome 3
Time Frame: Baseline, Day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 7 | 7 | 8
log IU/mL
  No Decrease: number analyzed (Participants) | 2 | 0 | 0
  No Decrease | 0.009 (0.010) |  |
  1 participant analyDecrease > 0 to < 0.5 log IU/mL: number analyzed (Participants) | 5 | 7 | 4
  1 participant analyDecrease > 0 to < 0.5 log IU/mL | -0.112 (0.147) | -0.171 (0.037) | -0.293 (0.112)
  Decrease 0.5 to 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 4
  Decrease 0.5 to 1.0 log IU/mL |  |  | -0.684 (0.179)
  Decrease > 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Test type: Superiority; p = 0.4615, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.0508, Fisher Exact
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.0769, Fisher Exact

9. Secondary Outcome: Change From Baseline at Day 99 in Log qHBsAg, by Category
Description: as for outcome 3
Time Frame: Baseline, Day 99
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 7 | 6 | 8
log IU/mL
  No Decrease: number analyzed (Participants) | 4 | 0 | 0
  No Decrease | 0.027 (0.018) |  |
  1 participant analyDecrease > 0 to < 0.5 log IU/mL: number analyzed (Participants) | 3 | 6 | 3
  1 participant analyDecrease > 0 to < 0.5 log IU/mL | -0.160 (0.202) | -0.210 (0.070) | -0.343 (0.110)
  Decrease 0.5 to 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 4
  Decrease 0.5 to 1.0 log IU/mL |  |  | -0.652 (0.068)
  Decrease > 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 1
  Decrease > 1.0 log IU/mL |  |  | -1.011 (NA) — 1 participant analyzed
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Test type: Superiority; p = 0.0699, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.0179, Fisher Exact
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.0430, Fisher Exact

10. Secondary Outcome: Change From Baseline at Day 113 in Log qHBsAg, by Category
Description: as for outcome 3
Time Frame: Baseline, Day 113
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 8
log IU/mL
  No Decrease: number analyzed (Participants) | 1 | 0 | 0
  No Decrease | 0.042 (NA) — 1 participant analyzed |  |
  1 participant analyDecrease > 0 to < 0.5 log IU/mL: number analyzed (Participants) | 5 | 6 | 4
  1 participant analyDecrease > 0 to < 0.5 log IU/mL | -0.115 (0.171) | -0.142 (0.045) | -0.359 (0.049)
  Decrease 0.5 to 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 4
  Decrease 0.5 to 1.0 log IU/mL |  |  | -0.726 (0.228)
  Decrease > 1.0 log IU/mL: number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ARC-520 1.0 mg/kg; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.0849, Fisher Exact
Statistical Analysis 3: Comparison: ARC-520 1.0 mg/kg vs ARC-520 2.0 mg/kg; Test type: Superiority; p = 0.0849, Fisher Exact

11. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths, and Discontinuations Due to AEs
Description: An AE is any untoward medical occurrence which does not necessarily have to have a causal relationship with this treatment. A treatment emergent AE (TEAE) was defined as an AE that was not present prior to the first study drug administration and started at/after the time of initiation of administration of study drug, or an AE which was present prior to initiation of study drug administration, which increased in severity after study drug administration. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a medically important event or reaction.
Time Frame: Through Day 169 (± 3 days)
Population: Safety Population: all participants who received at least one dose of study drug or placebo, and had at least one post-dose safety assessment.
Measure: Number; unit: participants
Arm/Group | Placebo Low Dose Comparator | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 6 | 5 | 10 | 11
participants
  ≥ 1 AE | 4 | 0 | 6 | 3
  ≥ 1 TEAE | 4 | 0 | 5 | 3
  ≥ 1 Serious TEAE | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0
  ≥ 1 TEAE Leading to Study Discontinuation | 0 | 0 | 0 | 0
  ≥ 1 TEAE Leading to Treatment Discontinuation | 0 | 0 | 0 | 0

12. Secondary Outcome: Pharmacokinetics of ARC-520: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: Due to the early suspension and termination of the study, all pharmacokinetic analyses were removed from the initial statistical analysis plan for this study. No collected samples were analyzed and all were destroyed.
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Pharmacokinetics of ARC-520: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Quantifiable Plasma Concentration (AUClast)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 12
Arm/Group | Placebo | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Pharmacokinetics of ARC-520: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 12
Groups:
- Placebo High Dose Comparator: Placebo (low dose or high dose comparator) once every 4 weeks for 4 doses, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day)
Arm/Group | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Pharmacokinetics of ARC-520: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 12
Arm/Group | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Pharmacokinetics of ARC-520: Clearance (CL)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 12
Arm/Group | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Pharmacokinetics of ARC-520: Apparent Volume of Distribution (V)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 12
Arm/Group | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Pharmacokinetics of ARC-520: Terminal Elimination Rate Constant (Kel)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 12
Arm/Group | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Pharmacokinetics of ARC-520: Terminal Elimination Half-Life (t1/2)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 12
Arm/Group | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through Day 169 (± 3 days)
Arm/Group | Placebo Low Dose Comparator | Placebo High Dose Comparator | ARC-520 1.0 mg/kg | ARC-520 2.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 4/6 | 0/5 | 5/10 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Low Dose Comparator (N=6) | Placebo High Dose Comparator (N=5) | ARC-520 1.0 mg/kg (N=10) | ARC-520 2.0 mg/kg (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No